CLINICAL TRIAL: NCT02589132
Title: Mobile-Thrive - A Family Self-Management Approach to Failure to Thrive
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Praveen Goday, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHW 15/22
Record Dates: First submitted 2015-09-03; First posted 2015-10-28 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Failure to Thrive
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Families receiving Standard of Care
- Mobile-Thrive application (Experimental): Standard care plus Mobile-Thrive app
  Interventions: Other: Mobile-Thrive application

INTERVENTIONS:
Other: Mobile-Thrive application — Families receive standard of care plus the Mobile-Thrive application
  Arms: Mobile-Thrive application

SUMMARY:
Failure to Thrive negatively affects growth, cognition, behavior, and quality of life (QoL), which can be devastating and enduring. These outcomes are high-cost and lead to increased family stress and negatively affect the caregiver-child relationship. Therefore, families need increased access to materials that will help them understand their child's health and help them use new feeding behaviors to improve the child's nutrition and growth. Standard care with the addition of Mobile Thrive (M-Thrive), our innovative smart phone-based mobile app, is intended to demonstrate the clinical advantages of using mobile health technology (mHealth) in comparison to standard care alone.

DETAILED DESCRIPTION:
Families will be randomly assigned to either the Standard Care plus access to the Mobile-Thrive (M-Thrive) application or Standard Care alone. All families will complete a 24-hour dietary recall, Feeding Strategies Questionnaire (FSQ), PedsQL Family Impact Module (PedsQL FIM), and Pediatric Inventory for Parents (PIP) at pre/post treatment. It will take about 45 minutes to complete these measures. Anthropometric measurements will be collected at pretreatment, 6 weeks, and 3 months. Families receiving standard care alone will have regularly scheduled visits in the Nutritional Care Program and will have access to standard care resources, including phone contacts and electronic access through the CHW hospital portal. Specifically, standard care treatment provides dietary and behavioral instructions on appropriate beverage intake, appropriate feeding regimen, advice on limiting low-calorie foods, and multivitamin supplementation, if appropriate. Families in the standard care plus the M-Thrive application will receive the standard care treatment that is described above, as well as on-demand resources, daily educational text messages, and family self-management push notifications through the M-Thrive application. The research team will train families on the use of the M-Thrive application and families in the standard care plus M-Thrive application can contact their provider through the application with questions and/or concerns. At the conclusion of the intervention, qualitative data regarding the participants' experience will be collected. Specifically, 90-minute focus group sessions will occur within 2 weeks of concluding the 3 month active phase of treatment. Families will be asked to discuss factors that affected their ability to sustain condition management recommendations, their efforts to access health care resources, factors that affect family quality of life and caregiver stress, and family impressions of what else would help to build support for families managing FTT. All sessions will be transcribed and coded for content analysis.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children ages 4 months to 4 years old with a medical diagnosis of failure to thrive.
* English speaking.

Exclusion Criteria:

* Parents of children who do not meet the inclusion criteria.
* Non- english speaking.

Ages: 4 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Weight z score | 3 months
  Change in weight as measured by weight z score percentiles

OTHER OUTCOMES:
Calorie intake | 3 months
  Change in calorie intake

CONTACTS AND LOCATIONS:
Overall Officials: Praveen Goday, MD, Principal Investigator — Medical College of Wisconsin; Alan Silverman, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Jaffe AC. Failure to thrive: current clinical concepts. Pediatr Rev. 2011 Mar;32(3):100-7; quiz 108. doi: 10.1542/pir.32-3-100. No abstract available. PMID 21364013
- [Background] Mitchell WG, Gorrell RW, Greenberg RA. Failure-to-thrive: a study in a primary care setting. Epidemiology and follow-up. Pediatrics. 1980 May;65(5):971-7. PMID 7367142
- [Background] Berwick DM, Levy JC, Kleinerman R. Failure to thrive: diagnostic yield of hospitalisation. Arch Dis Child. 1982 May;57(5):347-51. doi: 10.1136/adc.57.5.347. PMID 6807215
- [Background] Skuse DH. Non-organic failure to thrive: a reappraisal. Arch Dis Child. 1985 Feb;60(2):173-8. doi: 10.1136/adc.60.2.173. PMID 3883912
- [Background] Block RW, Krebs NF; American Academy of Pediatrics Committee on Child Abuse and Neglect; American Academy of Pediatrics Committee on Nutrition. Failure to thrive as a manifestation of child neglect. Pediatrics. 2005 Nov;116(5):1234-7. doi: 10.1542/peds.2005-2032. PMID 16264015
- [Background] Black MM, Krishnakumar A. Predicting longitudinal growth curves of height and weight using ecological factors for children with and without early growth deficiency. J Nutr. 1999 Feb;129(2S Suppl):539S-543S. doi: 10.1093/jn/129.2.539S. PMID 10064327
- [Background] Dowdney L, Skuse D, Morris K, Pickles A. Short normal children and environmental disadvantage: a longitudinal study of growth and cognitive development from 4 to 11 years. J Child Psychol Psychiatry. 1998 Oct;39(7):1017-29. PMID 9804034
- [Background] Dykman RA, Casey PH, Ackerman PT, McPherson WB. Behavioral and cognitive status in school-aged children with a history of failure to thrive during early childhood. Clin Pediatr (Phila). 2001 Feb;40(2):63-70. doi: 10.1177/000992280104000201. PMID 11261452
- [Background] Drotar D, Sturm L. Prediction of intellectual development in young children with early histories of nonorganic failure-to-thrive. J Pediatr Psychol. 1988 Jun;13(2):281-96. doi: 10.1093/jpepsy/13.2.281. No abstract available. PMID 3171820
- [Background] Skuse D, Pickles A, Wolke D, Reilly S. Postnatal growth and mental development: evidence for a "sensitive period". J Child Psychol Psychiatry. 1994 Mar;35(3):521-45. doi: 10.1111/j.1469-7610.1994.tb01738.x. PMID 7515070
- [Background] Mendez MA, Adair LS. Severity and timing of stunting in the first two years of life affect performance on cognitive tests in late childhood. J Nutr. 1999 Aug;129(8):1555-62. doi: 10.1093/jn/129.8.1555. PMID 10419990
- [Background] Yang S, Tilling K, Martin R, Davies N, Ben-Shlomo Y, Kramer MS. Pre-natal and post-natal growth trajectories and childhood cognitive ability and mental health. Int J Epidemiol. 2011 Oct;40(5):1215-26. doi: 10.1093/ije/dyr094. Epub 2011 Jul 15. PMID 21764769
- [Background] Crookston BT, Penny ME, Alder SC, Dickerson TT, Merrill RM, Stanford JB, Porucznik CA, Dearden KA. Children who recover from early stunting and children who are not stunted demonstrate similar levels of cognition. J Nutr. 2010 Nov;140(11):1996-2001. doi: 10.3945/jn.109.118927. Epub 2010 Sep 15. PMID 20844188
- [Background] Atalay A, McCord M. Characteristics of failure to thrive in a referral population: implications for treatment. Clin Pediatr (Phila). 2012 Mar;51(3):219-25. doi: 10.1177/0009922811421001. Epub 2011 Oct 12. PMID 21997145
- [Background] Garro A, Thurman SK, Kerwin ME, Ducette JP. Parent/caregiver stress during pediatric hospitalization for chronic feeding problems. J Pediatr Nurs. 2005 Aug;20(4):268-75. doi: 10.1016/j.pedn.2005.02.015. PMID 16030506
- [Background] Rumberger JS, Dansky K. Is there a business case for telehealth in home health agencies? Telemed J E Health. 2006 Apr;12(2):122-7. doi: 10.1089/tmj.2006.12.122. PMID 16620166
- [Background] Gazmararian JA, Elon L, Yang B, Graham M, Parker R. Text4baby program: an opportunity to reach underserved pregnant and postpartum women? Matern Child Health J. 2014 Jan;18(1):223-232. doi: 10.1007/s10995-013-1258-1. PMID 23494485
- [Background] Ryan P, Sawin KJ. The Individual and Family Self-Management Theory: background and perspectives on context, process, and outcomes. Nurs Outlook. 2009 Jul-Aug;57(4):217-225.e6. doi: 10.1016/j.outlook.2008.10.004. PMID 19631064
- [Background] Black MM, Dubowitz H, Hutcheson J, Berenson-Howard J, Starr RH Jr. A randomized clinical trial of home intervention for children with failure to thrive. Pediatrics. 1995 Jun;95(6):807-14. PMID 7539121
- [Background] Black MM, Dubowitz H, Krishnakumar A, Starr RH Jr. Early intervention and recovery among children with failure to thrive: follow-up at age 8. Pediatrics. 2007 Jul;120(1):59-69. doi: 10.1542/peds.2006-1657. PMID 17606562
- [Background] Hutcheson JJ, Black MM, Talley M, Dubowitz H, Howard JB, Starr RH Jr, Thompson BS. Risk status and home intervention among children with failure-to-thrive: follow-up at age 4. J Pediatr Psychol. 1997 Oct;22(5):651-68. doi: 10.1093/jpepsy/22.5.651. PMID 9383928
- [Background] Raynor P, Rudolf MC, Cooper K, Marchant P, Cottrell D. A randomised controlled trial of specialist health visitor intervention for failure to thrive. Arch Dis Child. 1999 Jun;80(6):500-6. doi: 10.1136/adc.80.6.500. PMID 10331996
- [Background] Wright CM, Callum J, Birks E, Jarvis S. Effect of community based management in failure to thrive: randomised controlled trial. BMJ. 1998 Aug 29;317(7158):571-4. doi: 10.1136/bmj.317.7158.571. PMID 9721113
- [Background] Rotheram-Borus MJ, Tomlinson M, Swendeman D, Lee A, Jones E. Standardized functions for smartphone applications: examples from maternal and child health. Int J Telemed Appl. 2012;2012:973237. doi: 10.1155/2012/973237. Epub 2012 Dec 13. PMID 23304136
- [Background] Klesges RC, Klesges LM, Brown G, Frank GC. Validation of the 24-hour dietary recall in preschool children. J Am Diet Assoc. 1987 Oct;87(10):1383-5. PMID 3655169
- [Background] Berlin KS, Davies WH, Silverman AH, Rudolph CD. Assessing family-based feeding strategies, strengths, and mealtime structure with the Feeding Strategies Questionnaire. J Pediatr Psychol. 2011 Jun;36(5):586-95. doi: 10.1093/jpepsy/jsp107. Epub 2009 Dec 7. PMID 19995867
- [Background] Davies WH, Satter E, Berlin KS, Sato AF, Silverman AH, Fischer EA, Arvedson JC, Rudolph CD. Reconceptualizing feeding and feeding disorders in interpersonal context: the case for a relational disorder. J Fam Psychol. 2006 Sep;20(3):409-17. doi: 10.1037/0893-3200.20.3.409. PMID 16937997
- [Background] Varni JW, Sherman SA, Burwinkle TM, Dickinson PE, Dixon P. The PedsQL Family Impact Module: preliminary reliability and validity. Health Qual Life Outcomes. 2004 Sep 27;2:55. doi: 10.1186/1477-7525-2-55. PMID 15450120
- [Background] Panepinto JA, Hoffmann RG, Pajewski NM. A psychometric evaluation of the PedsQL Family Impact Module in parents of children with sickle cell disease. Health Qual Life Outcomes. 2009 Apr 16;7:32. doi: 10.1186/1477-7525-7-32. PMID 19371442
- [Background] Streisand R, Braniecki S, Tercyak KP, Kazak AE. Childhood illness-related parenting stress: the pediatric inventory for parents. J Pediatr Psychol. 2001 Apr-May;26(3):155-62. doi: 10.1093/jpepsy/26.3.155. PMID 11259517